CLINICAL TRIAL: NCT00749268
Title: Evaluation of Postoperative Pain Following Laparoscopic Hernia Repair: A Prospective, Randomized Comparison to Evaluate the Incidence of Post-operative Pain Associated With Absorbable Fixation (AbsorbaTack) vs Conventional Fixation (ProTack) Following Laparoscopic Hernia Repair
Brief Title: AbsorbaTack Evaluation of Postoperative Pain Following Laparoscopic Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS08011
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Hernia, Inguinal; Hernia, Ventral
Keywords: hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Device: AbsorbaTack
- B (Active Comparator)
  Interventions: Device: ProTack

INTERVENTIONS:
Device: AbsorbaTack — Comparison of different devices for mesh fixation. This intervention arm has absorbable tacks as the method of hernia mesh fixation. Application is during hernia repair and tacks will essentially absorb within the body after 1 year.
  Arms: A
Device: ProTack — Comparison of different devices for mesh fixation. This intervention is a permanent tack for hernia mesh fixation. Application is during hernia repair and the tacks will remain in the body.
  Arms: B

SUMMARY:
The objective of this study is to assess pain that occurs following hernia repair that is related to mesh fixation. The study is designed to see if there is any difference in pain after surgery between absorbable and permanent methods of mesh fixation in inguinal and ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and comply with the schedule of protocol assessments
* Age > 18 years
* Subjects undergoing laparoscopic hernia repair with Parietex or Parietex Composite reinforcements depending on indication and fixation of reinforcements with helical tackers (ProTack, Covidien) or absorbable tacks (AbsorbaTack, Covidien) in accordance with recommendations for use

Exclusion Criteria:

* Pregnancy
* Patients considered to have greater than reasonable surgical risk associated with general anesthesia and laparoscopic hernia repair
* Known active infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics or oral antibiotics within 30 days prior to screening
* History of alcohol or drug abuse within 6 months prior to screening
* History of chronic pain condition requiring more than 30 days of medical management
* Use of an additional nonresorbable means of fixation (inguinal)
* Patients considered not able to comply with the protocol and follow up schedule
* ASA grade of 4 or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Rosen, Principal Investigator — Case Medical Center, University Hospitals of Cleveland, Cleveland, OH, USA
Locations (2):
- United States (2):
  - University Hospitals at Case Medical Center, Cleveland, Ohio
  - Greenville Hospital System, Greenville, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 4, 2008 and November 4, 2010, 117 subjects signed informed consent for the inguinal hernia arm of the study and 113 for the ventral arm. Of those subjects who consented, 106 and 110 were randomized to a treatment group (either AbsorbaTack™ or ProTack™) for inguinal and ventral hernia repair, respectively.
Groups:
- Inguinal Arm: Patients with inguinal hernias are randomized to receive either AbsorbaTack or ProTack. The two treatments are compared within a single hernia type but not across hernia types.
- Ventral Arm: Patients with ventral hernias are randomized to receive either AbsorbaTack or ProTack. The two treatments are compared within a single hernia type but not across hernia types.
Period: Overall Study
Arm/Group | Inguinal Arm | Ventral Arm
Started | 106 | 110
Completed | 72 | 74
Not Completed | 34 | 36

BASELINE CHARACTERISTICS:
Population: 1 inguinal pt assigned to receive AbsorbaTack was treated with ProTack and one patient assigned to receive ProTack received AbsorbaTack. These patients are included in the "intent to treat" population above, but were omitted from the safety population.
Groups:
- Inguinal Arm - AbsorbaTack: Inguinal hernia study arm with AbsorbaTack as treatment.
- Inguinal Arm - ProTack: Inguinal hernia study arm with ProTack as treatment.
- Ventral Arm - Absorbatack: Ventral hernia study arm with AbsorbaTack as treatment.
- Ventral Arm - ProTack: Ventral hernia study arm with ProTack as treatment.
- Total: Total of all reporting groups
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack | Total
Number analyzed (Participants) | 52 | 52 | 56 | 54 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (15.5) | 53.3 (12.3) | 50.3 (11.3) | 53.8 (12.9) | 51.49 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 20 | 27 | 55
  Male | 51 | 45 | 36 | 27 | 159
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 31 | 29 | 127
  France | 14 | 13 | 19 | 19 | 65
  Germany | 4 | 6 | 6 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Pain Intensity Numeric Rating Scale (PI-NRS) - change from baseline. Treatments analyzed within inguinal arm and within ventral arm.
  Scale is 0 - 10 with 0 being "no pain" and 10 being "worst pain imaginable".
Time Frame: Discharge, Month 1, Month 6, Month 12
Population: 1 patient in the Ventral Arm - AbsorbaTack had only pre-operative pain scores available so was unable to be included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack
Number analyzed (Participants) | 52 | 52 | 55 | 54
units on a scale
  Change from baseline - discharge | .8 (2.8) | 2.0 (2.2) | 2.2 (3.8) | 3.3 (3.6)
  Change from baseline - 1 month | -1.1 (2.7) | -.4 (1.8) | -.7 (3.0) | .5 (1.9)
  Change from baseline - 6 months | -1.8 (2.4) | -.6 (1.8) | -1.3 (2.8) | -.6 (1.7)
  Change from baseline - 1 year | -1.2 (2.3) | -.9 (1.6) | -1.8 (2.7) | -.8 (1.8)

2. Primary Outcome: Safety for Laparoscopic Hernia Repair as Measured by Number of Patients Experiencing Device Related Events
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack
Number analyzed (Participants) | 53 | 51 | 55 | 54
participants | 7 | 8 | 7 | 8

3. Secondary Outcome: Quality of Life
Description: Quality of life as measured by the SF-12 which is a multipurpose short form survey with 12 questions. The questions were combined, scored, and weighted to create a scale that provide glimpses into physical functioning and overall health-related-quality of life.
  The Physical Composite Score was computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Pre-op, Month 1, Month 6, 1 year
Population: Participant # above reflects those at pre-op. Arms ended study with 34, 39, 36 and 39 subjects, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack
Number analyzed (Participants) | 50 | 50 | 55 | 53
units on a scale
  Pre-Op | 48.8 (8.6) | 50.6 (8.1) | 46.1 (9.3) | 49.0 (9.1)
  1 Month | 49.1 (7.9) | 50.2 (7.0) | 45.4 (9.5) | 45.2 (9.0)
  6 Month | 55.3 (6.6) | 54.4 (6.3) | 51.6 (9.4) | 51.1 (7.6)
  1 year | 55.8 (7.4) | 53.8 (6.0) | 52.0 (8.1) | 53.3 (6.6)

4. Secondary Outcome: Hernia Recurrence
Time Frame: Discharge, 1 Month, 6 Month, 1 year
Measure: Number; unit: participants
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack
Number analyzed (Participants) | 52 | 52 | 56 | 54
participants
  Discharge | 0 | 1 | 0 | 0
  1 Month | 0 | 1 | 1 | 2
  6 Month | 2 | 1 | 3 | 0
  1 Year | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from time of randomization through 1 year.
Description: Inguinal Arm - 1 patient randomized to ProTack group was treated w/AbsorbaTack and 1 patient randomized to the AbsorbaTack group was treated w/ProTack, so these 2 patients were not included in the safety analysis set.
  Ventral Arm - 1 patient randomized to the AbsorbaTack group was treated w/ProTack so what not included in the safety analysis set
Arm/Group | Inguinal Arm - AbsorbaTack | Inguinal Arm - ProTack | Ventral Arm - Absorbatack | Ventral Arm - ProTack
Serious Adverse Events (participants affected / at risk) | 6/53 | 6/51 | 8/55 | 9/54
Other Adverse Events (participants affected / at risk) | 17/53 | 20/51 | 24/55 | 33/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inguinal Arm - AbsorbaTack (N=53) | Inguinal Arm - ProTack (N=51) | Ventral Arm - Absorbatack (N=55) | Ventral Arm - ProTack (N=54)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Oesophagectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Spinal laminectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Adrenocortical Insufficiency Acute (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Suture Related Complication (General disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laparotomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inguinal Arm - AbsorbaTack (N=53) | Inguinal Arm - ProTack (N=51) | Ventral Arm - Absorbatack (N=55) | Ventral Arm - ProTack (N=54)
Seroma (Injury, poisoning and procedural complications) | 9 | 12 | 13 | 19
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 4 | 4
Incision Site Pain (Injury, poisoning and procedural complications) | 5 | 2 | 3 | 3
Urinary Retention (Renal and urinary disorders) | 3 | 1 | 4 | 3
Haemorrhage (Vascular disorders) | 0 | 3 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less